CLINICAL TRIAL: NCT05282472
Title: Exercising With a Surgical Mask is Safe But Decreases Performance in Both Athletic and Non-athletic Individuals
Brief Title: Exercising With a Surgical Mask in Both Athletic and Non-athletic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şensu Dinçer (Other)
Responsible Party: Sponsor-Investigator, Şensu Dinçer, medical doctor, Istanbul University
Organization: Istanbul University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: Exercising with a mask
Record Dates: First submitted 2022-02-03; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: surgical mask; Cardiopulmonary exercise test; COVID-19 (coronovirus-19 disease); exercise
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: A prospective, crossover designed study was conducted in 2 phases. Cardiopulmonary exercise test was performed with and without surgical mask in all participants in between 48 hours. The participant group was further divided into two groups as athlete and non-athlete. In first step, parameters were compared between the CPET tests performed with and without surgical masks. In second step, athletes' and non-athletes' parameters were compared during CPET tests performed with surgical mask.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with surgical mask (Experimental): all participants who were applied CPET with surgical mask
  Interventions: Diagnostic Test: CPET with mask
- without surgical mask (Active Comparator): all participants who were applied CPET without surgical mask
  Interventions: Diagnostic Test: CPET without mask

INTERVENTIONS:
Diagnostic Test: CPET without mask — Regular cardiopulmonary exercise tests were applied to all participants in phase 1.
  Arms: without surgical mask
Diagnostic Test: CPET with mask — A 3-layer surgical mask was placed on CPET device's mask and was fixed with a CPET tribune. In phase 2, as using this combined (surgical mask and device's mask) masks, CPETs were performed in all participants again, after 48 hours.
  Arms: with surgical mask

SUMMARY:
This study aimed to examine the impact of surgical masks on maximal and submaximal exercise in both athlete and non-athlete individuals.

DETAILED DESCRIPTION:
All participants will be informed about the procedure and, will sign an informed consent form. They will undergone a detailed physical examination before enrollment in the study. The study is conducted in 2-phases, in non-randomized, controlled design. Cardiopulmonary exercise tests (CPET) are going to be performed with and without a surgical mask with 48 hours in between.

ELIGIBILITY:
Inclusion Criteria:

* healthy athletes
* healthy non-athletes

Exclusion Criteria:

* any musculoskeletal, cardiac or respiratory problem

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
maximum oxygen consumption (VO2max) change between CPET with surgical mask and without surgical mask | two CPET tests which will be carried out two days within 2 weeks
  Cardiopulmonary exercise test (CPET) is a well known, gold standard test to measure VO2 max during exercise. The higher VO2 max value shows better endurance.VO₂ max is the maximum (max) rate (V) of oxygen (O₂) the body is able to use during exercise
max minute ventilation (VEmax) change between CPET with surgical mask and without surgical mask | two CPET tests which will be carried out two days within 2 weeks
  VEmax is the maximum volume of gas inhaled (inhaled minute volume) or exhaled (exhaled minute volume) from a person's lungs per minute.
exercise test duration change between CPET with surgical mask and without surgical mask | two CPET tests which will be carried out two days within 2 weeks
  CPET duration of a participant
end-tidal carbon dioxide pressure (pETCO2) change at the maximum and anaerobic levels of CPET | two CPET tests which will be carried out two days within 2 weeks
  End-tidal carbon dioxide pressure (pETCO2) is the level of carbon dioxide that is released at the end of an exhaled breath.
End-tidal partial oxygen pressure (pETO2) change at the maximum and anaerobic levels of CPET | two CPET tests which will be carried out two days within 2 weeks
  refers to PO2 of exhaled gas. It is measured at the end of exhalation and its units are mm Hg.
Tidal volume (TV) change at the maximum and anaerobic levels of CPET | two CPET tests which will be carried out two days within 2 weeks
  TV that volume of air moved into or out of the lungs during quiet breathing

SECONDARY OUTCOMES:
minute ventilation at anerobic level (VEan) results of athlete and non-athlete comparison | 2 weeks
  The VEan difference in between the changes in CPETs with and without masks of athletes and non-athletes
maximum minute ventilation (VEmax) results of athlete and non-athlete comparison | 2 weeks
  The VEmax difference in between the changes in CPETs with and without masks of athletes and non-athletes
VO2max results of athlete and non-athlete comparison | 2 weeks
  The VO2max difference in between the changes in CPETs with and without masks of athletes and non-athletes
VO2an results of athlete and non-athlete comparison | 2 weeks
  The VO2an difference in between the changes in CPETs with and without masks of athletes and non-athletes
PETO2 results of athlete and non-athlete comparison | 2 weeks
  The PETO2 difference in between the changes in CPETs with and without masks of athletes and non-athletes
PETCO2 | 2 weeks
  The PETCO2 difference in between the changes in CPETs with and without masks of athletes and non-athletes

CONTACTS AND LOCATIONS:
Locations (1):
- Şensu Dinçer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD)that will underlie results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 1 year after publication
Access Criteria: IPD can be shared by researchers such as exercise physiologists, sports scientist and sport medicine physicians